CLINICAL TRIAL: NCT04075812
Title: High Definition Neuromuscular Stimulation in Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Marcia Bockbrader, Assistant Professor- Physical Medicine & Rehabilitation, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013H0092
Record Dates: First submitted 2019-01-31; First posted 2019-09-03 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-08

CONDITIONS: Spinal Cord Injury at C4-C6 Level
Keywords: reanimation; stimulation

STUDY DESIGN:
Intervention Model Description: Single arm, open-label, non-controlled prospective intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Neuromuscular Stimulator (Experimental): Neuromuscular Stimulator is setup and calibrated, various spatial and temporal stimulation patterns will be tested to evoke wrist/hand movements in various sequences of individual and combined movements.
  Interventions: Device: Neuromuscular Stimulator

INTERVENTIONS:
Device: Neuromuscular Stimulator

SUMMARY:
The purpose of this study is to demonstrate high definition non-invasive neuromuscular stimulation of an upper extremity in tetraplegic participants.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) is an insult to the spinal cord resulting in a change, either temporary or permanent, in its normal motor, sensory, and/or autonomic function. It is estimated that the annual incidence of spinal cord injury (SCI), not including those who die at the scene of the accident, is approximately 40 cases per million population in the U. S. or approximately 12,000 new cases each year.

The purpose of this study is to demonstrate high definition non-invasive neuromuscular stimulation of an upper extremity in tetraplegic participants. This study will plan to enroll up to 15 subjects who have been diagnosed with tetraplegia. The total duration of the study is expected to be about 18 months, and each participant is expected to be on the study for about 6 months.

The study design will consist of the following two (2) phases listed below. I. Baseline assessment and calibration (approximately 1 month) II. Testing motions: pre-sequenced and EEG-triggered motions; further calibration as needed (approximately 5 months)

Phase I - Baseline

* Medical history review
* Physical and neurological exam
* EMG
* Fit and calibrate external stimulator: The Battelle Neuromuscular Stimulator will be setup and calibrated to evoke wrist and hand/finger movements.

Phase II - Testing Motions After the Neuromuscular Stimulator is setup and calibrated, various spatial and temporal stimulation patterns will be tested to evoke wrist/hand movements in various sequences of individual and combined movements.

ELIGIBILITY:
Inclusion Criteria:

* Must be 21 years or older.

  * Must be tetraplegic (C4-6 ASIA A)
  * 12 months post injury and neurologically stable
  * Participant is willing to comply with all follow-up evaluations at the specified times.
  * Participant is able to provide informed consent prior to enrollment in the study.
  * The participant is fluent in English.

Exclusion Criteria:

* No active wound healing or skin breakdown issues.

  * No history of poorly controlled autonomic dysreflexia.
  * Other implantable devices such as heart/brain pacemakers
  * Subjects who rely on ventilators

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04-25 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Bockbrader, MD PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center - Center for Neuromodulation, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bouton CE, Shaikhouni A, Annetta NV, Bockbrader MA, Friedenberg DA, Nielson DM, Sharma G, Sederberg PB, Glenn BC, Mysiw WJ, Morgan AG, Deogaonkar M, Rezai AR. Restoring cortical control of functional movement in a human with quadriplegia. Nature. 2016 May 12;533(7602):247-50. doi: 10.1038/nature17435. Epub 2016 Apr 13. PMID 27074513
- [Background] Sharma G, Friedenberg DA, Annetta N, Glenn B, Bockbrader M, Majstorovic C, Domas S, Mysiw WJ, Rezai A, Bouton C. Using an Artificial Neural Bypass to Restore Cortical Control of Rhythmic Movements in a Human with Quadriplegia. Sci Rep. 2016 Sep 23;6:33807. doi: 10.1038/srep33807. PMID 27658585
- [Background] Friedenberg DA, Bouton CE, Annetta NV, Skomrock N, Mingming Zhang, Schwemmer M, Bockbrader MA, Mysiw WJ, Rezai AR, Bresler HS, Sharma G. Big data challenges in decoding cortical activity in a human with quadriplegia to inform a brain computer interface. Annu Int Conf IEEE Eng Med Biol Soc. 2016 Aug;2016:3084-3087. doi: 10.1109/EMBC.2016.7591381. PMID 28268963
- [Background] Friedenberg DA, Schwemmer MA, Landgraf AJ, Annetta NV, Bockbrader MA, Bouton CE, Zhang M, Rezai AR, Mysiw WJ, Bresler HS, Sharma G. Neuroprosthetic-enabled control of graded arm muscle contraction in a paralyzed human. Sci Rep. 2017 Aug 21;7(1):8386. doi: 10.1038/s41598-017-08120-9. PMID 28827605
- [Background] Colachis SC 4th, Bockbrader MA, Zhang M, Friedenberg DA, Annetta NV, Schwemmer MA, Skomrock ND, Mysiw WJ, Rezai AR, Bresler HS, Sharma G. Dexterous Control of Seven Functional Hand Movements Using Cortically-Controlled Transcutaneous Muscle Stimulation in a Person With Tetraplegia. Front Neurosci. 2018 Apr 4;12:208. doi: 10.3389/fnins.2018.00208. eCollection 2018. PMID 29670506
- [Background] Schwemmer MA, Skomrock ND, Sederberg PB, Ting JE, Sharma G, Bockbrader MA, Friedenberg DA. Meeting brain-computer interface user performance expectations using a deep neural network decoding framework. Nat Med. 2018 Nov;24(11):1669-1676. doi: 10.1038/s41591-018-0171-y. Epub 2018 Sep 24. PMID 30250141
- [Background] Skomrock ND, Schwemmer MA, Ting JE, Trivedi HR, Sharma G, Bockbrader MA, Friedenberg DA. A Characterization of Brain-Computer Interface Performance Trade-Offs Using Support Vector Machines and Deep Neural Networks to Decode Movement Intent. Front Neurosci. 2018 Oct 24;12:763. doi: 10.3389/fnins.2018.00763. eCollection 2018. PMID 30459542
- [Background] Bockbrader M, Annetta N, Friedenberg D, Schwemmer M, Skomrock N, Colachis S 4th, Zhang M, Bouton C, Rezai A, Sharma G, Mysiw WJ. Clinically Significant Gains in Skillful Grasp Coordination by an Individual With Tetraplegia Using an Implanted Brain-Computer Interface With Forearm Transcutaneous Muscle Stimulation. Arch Phys Med Rehabil. 2019 Jul;100(7):1201-1217. doi: 10.1016/j.apmr.2018.07.445. Epub 2019 Mar 20. PMID 30902630
- [Result] Annetta NV, Friend J, Schimmoeller A, Buck VS, Friedenberg DA, Bouton CE, Bockbrader MA, Ganzer PD, Colachis Iv SC, Zhang M, Mysiw WJ, Rezai AR, Sharma G. A High Definition Noninvasive Neuromuscular Electrical Stimulation System for Cortical Control of Combinatorial Rotary Hand Movements in a Human With Tetraplegia. IEEE Trans Biomed Eng. 2019 Apr;66(4):910-919. doi: 10.1109/TBME.2018.2864104. Epub 2018 Aug 7. PMID 30106673

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from Tertiary Care Center
Groups:
- Neuromuscular Stimulator: Neuromuscular Stimulator is setup and calibrated, various spatial and temporal stimulation patterns will be tested to evoke wrist/hand movements in various sequences of individual and combined movements.
  Neuromuscular Stimulator
Period: Overall Study
Arm/Group | Neuromuscular Stimulator
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neuromuscular Stimulator
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 31 [21 to 41]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Voluntary Movement
Description: consistent and repetitive voluntary movement in the targeted muscle groups as assessed by investigator(s)- no formal scale is used.
  The participant(s) started out with paralysis due to spinal cord injury, so any active voluntary movement consists of a qualitative change in movement.
Time Frame: through study completion, up to 60 months
Population: All enrolled patients were able to generate consistent and repetitive movement in targeted muscle groups
Measure: Count of Participants; unit: Participants
Arm/Group | Neuromuscular Stimulator
Number analyzed (Participants) | 2
Participants
  Evoked movement - able | 2
  Evoked movement - unable | 0

2. Secondary Outcome: Change in Functional Movement
Description: consistent movement in the targeted muscle groups that is functional (manipulate or pick up an object); as assessed by investigator(s) for task completion- no formal scale used Objects were taken from the Action Research Arm Task, Grasp and Release Task, GRASSP as well as using household objects (phone, cup, spoon)
Time Frame: through study completion, up to 60 months
Population: Consistent functional movement for object manipulation
Measure: Count of Participants; unit: Participants
Arm/Group | Neuromuscular Stimulator
Number analyzed (Participants) | 2
Participants
  Evoked object manipulation - able | 2
  Evoked object manipulation - unable | 0

ADVERSE EVENTS:
Time Frame: from baseline through study completion, up to 60 months
Description: Per clinicaltrials.gov definitions
Arm/Group | Neuromuscular Stimulator
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuromuscular Stimulator (N=2)
Device-related SAE (anticipated) (Skin and subcutaneous tissue disorders) | 1 (1) — Skin irritation/burns
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuromuscular Stimulator (N=2)
Non-device related AE associated with spinal cord injury (anticipated) (Renal and urinary disorders) | 2 (2) — Urinary tract infections and/or stones associated with neurogenic bladder
Non-device related AE associated with spinal cord injury (anticipated) (Skin and subcutaneous tissue disorders) | 1 (2) — Deep tissue injury complications

LIMITATIONS AND CAVEATS:
Both participants were in the chronic phase of their spinal cord injury. Muscle conditioning with neuromuscular stimulation was required for several weeks before functional object manipulation was observed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-01-31): https://cdn.clinicaltrials.gov/large-docs/12/NCT04075812/Prot_SAP_000.pdf